CLINICAL TRIAL: NCT01888120
Title: Patient Registry of Intrathecal Ziconotide Management (PRIZM): An Open-Label, Long Term, Multi-Center, Observational Study of PRIALT® (Ziconotide) Solution, Intrathecal Infusion, in Patients With Severe Chronic Pain
Brief Title: Patient Registry of Intrathecal Ziconotide Management(PRIZM)
Acronym: PRIZM
Status: Completed | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-001
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Patients With Severe Chronic Pain
MeSH Terms: interventions — ziconotide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe Chronic Pain
  Interventions: Drug: Ziconotide

INTERVENTIONS:
Drug: Ziconotide

SUMMARY:
The objectives of this study are to evaluate the effectiveness, long-term safety, tolerability, satisfaction with treatment, and health-related quality of life (HRQoL) associated with Intrathecal PRIALT use for severe chronic pain of varying etiologies.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age at the time of study entry.
* Patient who has severe chronic pain, whom IT therapy is warranted, and who is intolerant of, or refractory to other treatments, such as systemic analgesics, adjunctive therapies, and/or IT morphine.
* Patient is planned to be initiated on IT PRIALT as the sole agent in the pump at a participated site.
* Patient has not received PRIALT treatment administered continuously via Medtronic SynchroMed® II pump within the past 30 days.
* Patient has a life expectancy >6 months as determined by the physician.
* Patient is able to read, understand, and voluntarily sign the IRB-approved informed consent document prior to the performance of any study-specific procedures.
* Patient is able to understand and complete required assessments.

Exclusion Criteria:

* Patient has a known hypersensitivity to PRIALT or any of its formulation components.
* Patient has a pre-existing history of psychosis.
* Patient has infection at the microinjection site, uncontrolled bleeding diathesis, or known spinal canal obstruction that impairs circulation of cerebrospinal fluid.
* Patient is being initiated with PRIALT in conjunction with other IT agents.
* Patients with any other concomitant treatment or medical condition that, in the opinion of the clinician, would render IT administration hazardous.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 140 patients will be enrolled at approximatley 50 sites in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2013-07; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The effectiveness of PRIALT therapy for the management of severe chronic pain as evidenced by change in patient-reported pain intensity from baseline to 12 weeks after enrollment | 12 Weeks

SECONDARY OUTCOMES:
Evaluate the following from the patient's perspective via patient reported outcomes (PROs) | From week 12, every 3 months up to month 18
Evaluate the patient's global impression of change (PGIC) with PRIALT treatment | From week 12, every 3 months up to month 18
Evaluate changes in concomitant pain medication use | From week 12, every 3 months up to month 18
Evaluate long-term safety and tolerability data, including incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | From week 12, every 3 months up to month 18
The use of PRIALT in current clinical practice including dose at initiation, titration speed, effective dose, duration of treatment effect, use of other pain medications, etc. | From week 12, every 3 months up to month 18

CONTACTS AND LOCATIONS:
Overall Officials: I-Zu Huang, MD, Study Director — Jazz Pharmaceuticals
Locations (43):
- United States (43):
  - Tennessee Valley Pain Consultants, Huntsville, Alabama
  - Valley Pain Specialists, Chandler, Arizona
  - Desert Pain Institute, Mesa, Arizona
  - Valley Pain Specialists, Scottsdale, Arizona
  - White River Health System, Batesville, Arkansas
  - United Pain Care, Sherwood, Arkansas
  - Coastal Pain Research, Carlsbad, California
  - Pain Therapy Solutions, Chino, California
  - Pain Medicine Associates, Inc., Fountain Valley, California
  - University of California, San Diego, La Jolla, California
  - Napa Pain Institute, Napa, California
  - Cypress Ambulatory Surgery Center, Santa Maria, California
  - Orthopedic Pain Specialists, Santa Monica, California
  - Colorado Pain Clinic, Loveland, Colorado
  - St. Francis Pain Center, Wilmington, Delaware
  - Clearwater Pain Management, Clearwater, Florida
  - Florida Pain Institute, Merritt Island, Florida
  - AMPM Research Clinic, Miami, Florida
  - Kennedy-White Orthopaedic Center, Sarasota, Florida
  - JM Clinical Research, South Miami, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Shepherd Center, Inc, Atlanta, Georgia
  - Exodus Pain Clinic, Boise, Idaho
  - Thompson and Chou Center for PM&R, Louisville, Kentucky
  - Ana Pain Management, Clinton Township, Michigan
  - Kozmary Center for Pain Management, Las Vegas, Nevada
  - Spinal & Skeletal Pain Medicine, Utica, New York
  - The Center for Clinical Research/Carolinas Pain Institute, Winston-Salem, North Carolina
  - Integrated Pain Solutions, Columbus, Ohio
  - Summa Health System Western Reserve Hospital, Cuyahoga Falls, Ohio
  - Ashland Neurosurgery, Ashland, Oregon
  - Cedar Sinai Medical Center, Ashland, Oregon
  - OAG Interventional Pain Consultants, Portland, Oregon
  - Oregon Anesthesiologist Group Interventional Pain Consultants, Portland, Oregon
  - Einstein Physician Practice, Inc., Elkins Park, Pennsylvania
  - DNA Advanced Pain Treatment Center, Greensburg, Pennsylvania
  - Houston Pain Associates, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Space City Pain Specialists LLP, Webster, Texas
  - Advanced Spine and Pain, Stafford, Virginia
  - The Center for Pain Relief, Charleston, West Virginia
  - The Center of Pain Relief Tri-State, Huntington, West Virginia
  - Anesthesia & Chronic Pain / University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] McDowell GC, Saulino MF, Wallace M, Grigsby EJ, Rauck RL, Kim P, Vanhove GF, Ryan R, Huang IZ, Deer T. Effectiveness and Safety of Intrathecal Ziconotide: Final Results of the Patient Registry of Intrathecal Ziconotide Management (PRIZM). Pain Med. 2020 Nov 1;21(11):2925-2938. doi: 10.1093/pm/pnaa115. PMID 32472137
- [Derived] Deer T, Rauck RL, Kim P, Saulino MF, Wallace M, Grigsby EJ, Huang IZ, Mori F, Vanhove GF, McDowell GC 2nd. Effectiveness and Safety of Intrathecal Ziconotide: Interim Analysis of the Patient Registry of Intrathecal Ziconotide Management (PRIZM). Pain Pract. 2018 Feb;18(2):230-238. doi: 10.1111/papr.12599. Epub 2017 Jul 14. PMID 28449352